CLINICAL TRIAL: NCT00625365
Title: CARES (Contrast EchocArdiography REgistry for Safety Surveillance): A Prospective, Phase IV, Open-Label, Nonrandomized, Multicenter, Surveillance Registry Study to Evaluate the Safety of DEFINITY® in Clinical Practice
Brief Title: A Prospective, Phase IV, Surveillance Registry Study to Evaluate the Safety of DEFINITY® in Clinical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DMP 115-415
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2011-08

CONDITIONS: Cardiovascular Disease
Keywords: DEFINITY; Safety; Survelliance
MeSH Terms: conditions — Cardiovascular Diseases | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DEFINITY® (Perflutren Lipid Microsphere) (Other): Patients who had undergone unenhanced echocardiography yielding suboptimal images and who were determined by the Principal Investigator to require DEFINITY-enhanced echocardiography
  Interventions: Drug: DEFINITY®

INTERVENTIONS:
Drug: DEFINITY® — DEFINITY may be injected by either an intravenous or bolus injection or infusion. Dosage as per standard clinical practice and Package Insert
  Other Names: DEFINITY; Perflutren Lipid Microsphere injectable suspension

SUMMARY:
The purpose of this registry study is to gather safety information on the current clinical use of and the safety of DEFINITY®

ELIGIBILITY:
Inclusion criteria

* Patients who, in the investigator's opinion, require DEFINITY® echocardiography due to suboptimal, unenhanced images.

Exclusion criteria

* Known hypersensitivity to perflutren, DEFINITY®, or other echo contrast agent.
* Prior SAE associated with perflutren, DEFINITY®, or administration of other echo contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lee, MD, Study Director — Lantheus Medical Imaging
Locations (16):
- United States (16):
  - UCSD Medical Center, San Diego, California
  - Alfieri Cardiology, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Maine Research Associates, Auburn, Maine
  - Park Nicolett Institute, Saint Louis Park, Minnesota
  - Cardiovascular Consultants, P.C., Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - St. Luke's-Roosevelt Hospital, New York, New York
  - Mt Sinai Medical Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Heart Center Cardiology, Fargo, North Dakota
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Consultants in Cardiology, Fort Worth, Texas
  - University of Texas Medical Center, Galveston, Texas
  - The Methodist DeBakey Heart Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from hospitals and clinics in the USA between February 2008 and April 2009
Pre-assignment Details: There were no pre-assignment requirements for this study
Groups:
- DEFINITY®: Patients who had undergone unenhanced echocardiography yielding suboptimal images and who were determined by the Principal Investigator to require DEFINITY-enhanced echocardiography
Period: Overall Study
Arm/Group | DEFINITY®
Started | 1060
Completed | 1053 (Participants who were analyzed for safety)
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — No IV access | 5
Not completed — VSD | 1

BASELINE CHARACTERISTICS:
Groups:
- DEFINITY (Perflutren Lipid Microsphere): Patients who had undergone unenhanced echocardiography yielding suboptimal images and who were determined by the Principal Investigator to require DEFINITY-enhanced echocardiography
Arm/Group | DEFINITY (Perflutren Lipid Microsphere)
Number analyzed (Participants) | 1053
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 609
  >=65 years | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400
  Male | 653

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients With Death or Life Threatening Cardiopulmonary Events Occurring Following Definity Administration
Time Frame: during or within 30 minutes of administration
Population: The safety population was analyzed per the protocol
Measure: Number; unit: Participants
Arm/Group | DEFINITY®
Number analyzed (Participants) | 1053
Participants | 0

2. Secondary Outcome: Serious Adverse Events
Description: Summary of the number and percentage of participants with serious adverse events occuring following completion of DEFINITY administration
Time Frame: Through 24 hours
Measure: Number; unit: Participants
Arm/Group | DEFINITY®
Number analyzed (Participants) | 1053
Participants | 0

3. Secondary Outcome: Adverse Events
Description: Summary of the number and percentage of participants with adverse events occuring following completion of DEFINITY administration
Time Frame: Through 24 hours
Measure: Number; unit: Participants
Arm/Group | DEFINITY®
Number analyzed (Participants) | 1053
Participants | 114

ADVERSE EVENTS:
Time Frame: Through 24 hours post last dose
Arm/Group | DEFINITY®
Serious Adverse Events (participants affected / at risk) | 0/1053
Other Adverse Events (participants affected / at risk) | 35/1053
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEFINITY® (N=1053)
Nausea (Gastrointestinal disorders) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 13 (13)
Tremor (Nervous system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No